CLINICAL TRIAL: NCT02385396
Title: Evaluation Concerning the Influence of Myo-inositol Therapy on the Dynamics of Embryo Development in Patients Suffering From PCOS Undergoing ICSI Treatment
Brief Title: Myo-inositol Therapy on the Dynamics of Embryo Development in Patients Suffering From PCOS Undergoing ICSI Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Artur Wdowiak, MD PhD, Medical University of Lublin
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUL024
Record Dates: First submitted 2015-02-12; First posted 2015-03-11 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-03

CONDITIONS: Polycystic Ovary Syndrome; Infertility
Keywords: Polycystic Ovary Syndrome; Infertility; Myo-inositol; Intracytoplasmic sperm injection
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility | interventions — Folic Acid

ARMS (3):
- Group I (Placebo Comparator): 60 patients diagnosed with PCOS, not myo-inositol treated undergoing ICSI
- Group II (Experimental): 52 patients diagnosed with PCOS undergoing ICSI, taking Inofolic (myo-inositol + folic acid)
  Interventions: Dietary Supplement: Inofolic: myo-inositol and folic acid
- Group III (Placebo Comparator): 105 patients not diagnosed with PCOS undergoing ICSI, not taking myo-inositol

INTERVENTIONS:
Dietary Supplement: Inofolic: myo-inositol and folic acid — 4000 mg of myo-inositol and 0,4 mg of folic acid for 3 months preceding the ICSI procedure
  Arms: Group II

SUMMARY:
The purpose of this study is to analyse the activity of myo-inositol on pregnancy rate, embryo development dynamics and oestradiol and progesterone concentration in blood serum and Superoxide Dismutase (SOD) and catalase concentration in follicular fluid of patients with Polycystic Ovary Syndrome (PCOS) undergoing Intracytoplasmic Sperm Injection (ICSI).

ELIGIBILITY:
Inclusion Criteria:

ICSI treatment due to infertility

PCOS patients enrolled according to the criteria established by representatives of the American Society of Reproductive Medicine (ASRM) and the European Society of Human Reproduction and Embryology (ESHRE)

Exclusion Criteria:

Severe endometriosis BMI <17 and >30 Metabolic diseases Lowered ovarian reserve

Ages: 27 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 217 (Actual)
Dates: Primary Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Oestradiol (E2) level in blood serum (pg/ml) | Between 11th and 19th day of cycle, when the largest of the oocyte in the evaluation of ultrasound exceeded 17mm diameter,
Progesterone (ng/ml) level in blood serum | Between 11th and 19th day of cycle, when the largest of the oocyte in the evaluation of ultrasound exceeded 17mm diameter
Superoxide dismutase (SOD) activity level in follicular fluid (mIU/mg) | On puncture day or on collection day of oocytes, in practice, between 11th and 19th day of cycle
  The decision was taken when three conditions are met: the biggest oocyte exceeds 17mm, the endometrium was over 9mm (two layers) and estradiol level was greater than 150
Catalase activity level in follicular fluid (mIU/mg) | On puncture day or on collection day of oocytes, in practice, between 11th and 19th day of cycle
  The decision was taken when three conditions are met: the biggest oocyte exceeds 17mm, the endometrium was over 9mm (two layers) and estradiol level was greater than 150

SECONDARY OUTCOMES:
Period of blastocyst and embryo development | From the moment of puncture, between the 11th and 19th day of the cycle, for a maximum of seven days
  Embryo culture was evaluated by means of constant monitoring performed in 10-minute intervals with a camera placed inside the incubator.The t0 time was described as the hour of the ICSI. tF was defined as the first moment when pronuclei were already visible, whereas tC as the last moment of their visibility. The moment when a single cell embryo appeared after syngamy was determined as t1, and then the superseding divisions were marked as t2, t3, t4, t5, t6, t7, t8. tM stood for the beginning of morula formation, whereas tB was the time during which the first signs of blastocyst cavity could be seen.
Pregnancy rate | During the 7th week of pregnancy
  Ultrasound examination of the echo of the embryo and heart rate

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Lublin, Lublin, Lublin Voivodeship, Poland

REFERENCES:
- [Background] Aanesen A, Westerbotn M. Prospective study of a Swedish infertile cohort 2005-08: population characteristics, treatments and pregnancy rates. Fam Pract. 2014 Jun;31(3):290-7. doi: 10.1093/fampra/cmu003. Epub 2014 Mar 3. PMID 24591683
- [Background] Shorakae S, Boyle J, Teede H. Polycystic ovary syndrome: a common hormonal condition with major metabolic sequelae that physicians should know about. Intern Med J. 2014 Aug;44(8):720-6. doi: 10.1111/imj.12495. PMID 24909750
- [Background] Huang JY, Rosenwaks Z. In vitro fertilisation treatment and factors affecting success. Best Pract Res Clin Obstet Gynaecol. 2012 Dec;26(6):777-88. doi: 10.1016/j.bpobgyn.2012.08.017. Epub 2012 Oct 9. PMID 23059403
- [Background] Gougeon A. Regulation of ovarian follicular development in primates: facts and hypotheses. Endocr Rev. 1996 Apr;17(2):121-55. doi: 10.1210/edrv-17-2-121. No abstract available. PMID 8706629
- [Background] Seleem AK, El Refaeey AA, Shaalan D, Sherbiny Y, Badawy A. Superoxide dismutase in polycystic ovary syndrome patients undergoing intracytoplasmic sperm injection. J Assist Reprod Genet. 2014 Apr;31(4):499-504. doi: 10.1007/s10815-014-0190-7. Epub 2014 Feb 14. PMID 24526356
- [Background] Combelles CM, Holick EA, Racowsky C. Release of superoxide dismutase-1 by day 3 embryos of varying quality and implantation potential. J Assist Reprod Genet. 2012 Apr;29(4):305-11. doi: 10.1007/s10815-012-9711-4. Epub 2012 Jan 25. PMID 22274808
- [Background] Jakimiuk AJ, Szamatowicz J. [The role of inositol deficiency in the etiology of polycystic ovary syndrome disorders]. Ginekol Pol. 2014 Jan;85(1):54-7. doi: 10.17772/gp/1691. Polish. PMID 24505965
- [Background] Krepelka P. [Myo-inositol in the treatment of polycystic ovary syndrome]. Ceska Gynekol. 2014 Jun;79(3):242-6. Czech. PMID 25054962
- [Background] Chiu TT, Rogers MS, Law EL, Briton-Jones CM, Cheung LP, Haines CJ. Follicular fluid and serum concentrations of myo-inositol in patients undergoing IVF: relationship with oocyte quality. Hum Reprod. 2002 Jun;17(6):1591-6. doi: 10.1093/humrep/17.6.1591. PMID 12042283
- [Background] Papaleo E, Unfer V, Baillargeon JP, Fusi F, Occhi F, De Santis L. RETRACTED: Myo-inositol may improve oocyte quality in intracytoplasmic sperm injection cycles. A prospective, controlled, randomized trial. Fertil Steril. 2009 May;91(5):1750-1754. doi: 10.1016/j.fertnstert.2008.01.088. Epub 2008 May 7. PMID 18462730
- [Background] Gerli S, Mignosa M, Di Renzo GC. Effects of inositol on ovarian function and metabolic factors in women with PCOS: a randomized double blind placebo-controlled trial. Eur Rev Med Pharmacol Sci. 2003 Nov-Dec;7(6):151-9. PMID 15206484
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome. Fertil Steril. 2004 Jan;81(1):19-25. doi: 10.1016/j.fertnstert.2003.10.004. PMID 14711538
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS consensus workshop group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome (PCOS). Hum Reprod. 2004 Jan;19(1):41-7. doi: 10.1093/humrep/deh098. PMID 14688154
- [Result] Agarwal A, Aponte-Mellado A, Premkumar BJ, Shaman A, Gupta S. The effects of oxidative stress on female reproduction: a review. Reprod Biol Endocrinol. 2012 Jun 29;10:49. doi: 10.1186/1477-7827-10-49. PMID 22748101
- [Result] Bausenwein J, Serke H, Eberle K, Hirrlinger J, Jogschies P, Hmeidan FA, Blumenauer V, Spanel-Borowski K. Elevated levels of oxidized low-density lipoprotein and of catalase activity in follicular fluid of obese women. Mol Hum Reprod. 2010 Feb;16(2):117-24. doi: 10.1093/molehr/gap078. Epub 2009 Sep 3. PMID 19729414
- [Result] Nel-Themaat L, Nagy ZP. A review of the promises and pitfalls of oocyte and embryo metabolomics. Placenta. 2011 Sep;32 Suppl 3:S257-63. doi: 10.1016/j.placenta.2011.05.011. Epub 2011 Jun 23. PMID 21703683
- [Result] Kurus M, Karakaya C, Karalok MH, To G, Johnson J. The control of oocyte survival by intrinsic and extrinsic factors. Adv Exp Med Biol. 2013;761:7-18. doi: 10.1007/978-1-4614-8214-7_2. PMID 24097378
- [Result] Ashwood-Smith MJ, Edwards RG. DNA repair by oocytes. Mol Hum Reprod. 1996 Jan;2(1):46-51. doi: 10.1093/molehr/2.1.46. PMID 9238657
- [Result] Inbar-Feigenberg M, Choufani S, Butcher DT, Roifman M, Weksberg R. Basic concepts of epigenetics. Fertil Steril. 2013 Mar 1;99(3):607-15. doi: 10.1016/j.fertnstert.2013.01.117. Epub 2013 Jan 26. PMID 23357459
- [Result] Whitelaw N, Bhattacharya S, Hoad G, Horgan GW, Hamilton M, Haggarty P. Epigenetic status in the offspring of spontaneous and assisted conception. Hum Reprod. 2014 Jul;29(7):1452-8. doi: 10.1093/humrep/deu094. Epub 2014 May 8. PMID 24812310
- [Result] Azzarello A, Hoest T, Mikkelsen AL. The impact of pronuclei morphology and dynamicity on live birth outcome after time-lapse culture. Hum Reprod. 2012 Sep;27(9):2649-57. doi: 10.1093/humrep/des210. Epub 2012 Jun 26. PMID 22740496
- [Result] Kirkegaard K, Kesmodel US, Hindkjaer JJ, Ingerslev HJ. Time-lapse parameters as predictors of blastocyst development and pregnancy outcome in embryos from good prognosis patients: a prospective cohort study. Hum Reprod. 2013 Oct;28(10):2643-51. doi: 10.1093/humrep/det300. Epub 2013 Jul 30. PMID 23900207
- [Result] Gawecka JE, Marh J, Ortega M, Yamauchi Y, Ward MA, Ward WS. Mouse zygotes respond to severe sperm DNA damage by delaying paternal DNA replication and embryonic development. PLoS One. 2013;8(2):e56385. doi: 10.1371/journal.pone.0056385. Epub 2013 Feb 19. PMID 23431372
- [Result] Campbell A, Fishel S, Bowman N, Duffy S, Sedler M, Hickman CF. Modelling a risk classification of aneuploidy in human embryos using non-invasive morphokinetics. Reprod Biomed Online. 2013 May;26(5):477-85. doi: 10.1016/j.rbmo.2013.02.006. Epub 2013 Feb 19. PMID 23518033
- [Result] Bidzinska-Speichert B, Lenarcik A, Tworowska-Bardzinska U, Slezak R, Bednarek-Tupikowska G, Milewicz A, Krepula K. Pro12Ala PPAR gamma2 gene polymorphism in women with polycystic ovary syndrome. Ginekol Pol. 2011 Jun;82(6):426-9. PMID 21853931
- [Result] Carbone MC, Tatone C, Delle Monache S, Marci R, Caserta D, Colonna R, Amicarelli F. Antioxidant enzymatic defences in human follicular fluid: characterization and age-dependent changes. Mol Hum Reprod. 2003 Nov;9(11):639-43. doi: 10.1093/molehr/gag090. PMID 14561807
- [Result] Munoz M, Cruz M, Humaidan P, Garrido N, Perez-Cano I, Meseguer M. Dose of recombinant FSH and oestradiol concentration on day of HCG affect embryo development kinetics. Reprod Biomed Online. 2012 Oct;25(4):382-9. doi: 10.1016/j.rbmo.2012.06.016. Epub 2012 Jul 4. PMID 22877941